CLINICAL TRIAL: NCT02024776
Title: The Effectiveness of Tailored Physical Training Intervention (Prehabilitation) in High-risk Patients Underwent Major Abdominal Surgery on Postoperative Complications: Randomized Controlled Trial
Brief Title: Effectiveness of Prehabilitation Program for High-risk Patients Underwent Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Graciela Martinez-Palli, MD, PhD, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI13/00425; PI13/00425 (Other Grant/Funding Number: Instituto de Salud Carlos III)
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Abdominal Surgical Patient; High-risk Patient
Keywords: Training; Wellness; Aerobic capacity; Information and communication technology, surgical risk; Abdominal surgery
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehabilitation (Active Comparator): Prehabilitation program is defined as a tailored physical exercise program to be carried out to a patient on the basis of his/her health condition, social circumstances and adherence profile. The intervention consisted of a standard 4-6 week supervised outpatient program including global endurance exercise training, or educational sessions followed by a self-management program supported by ICT during the follow-up period, or a combination of both.
  Interventions: Behavioral: Prehabilitation
- No-intervention (No Intervention): Standard counseling and conventional pre-surgical measures

INTERVENTIONS:
Behavioral: Prehabilitation — Tailored exercise training program
  Arms: Prehabilitation

SUMMARY:
Despite recent advances, morbidity and mortality associated to major abdominal surgery is significant. A poor physical condition and functional status reduces the ability of a person to cope, mentally and physically, with hospitalization and surgery and may compromise functional recovery, potentially leading to postoperative complications and death. Prehabilitation aims to enhance functional capacity preoperatively for better toleration of surgery and to facilitate recovery and eventually the prognosis of the surgical patient. Whereas the benefits of cardiopulmonary fitness programs are well established, the accessibility, sustainability of effects, and impact on the surgical outcome of these programs are unsolved issues. Wellness programs based on integrated care services supported by Information and Communication Technology (ICT) can overcome such limitations. The investigators hypothesized that a prehabilitation program, inducing beneficial effects on exercise capacity, may improve the surgical outcome in high-risk patients. Moreover, ICT support may contribute to increase the adherence and sustainability of this intervention.

ELIGIBILITY:
Inclusion Criteria:

Patients over 70 years-old and/or American Society of Anesthesiologists (ASA) health status class III-IV, with a DASI (Duke Activity Score Index) <46 points, referred for scheduled major abdominal surgery

Exclusion Criteria:

* Unstable severe co-morbid disease
* Dementia and psychosis, severe mental disorder or substance abuse or dependence
* Disabling orthopedic and neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative complications, classified by Clavien Scale | Time Frame: 30days or the postoperative hospital stay if longer than 30 days

SECONDARY OUTCOMES:
Length of stay | 30 days or the postoperative hospital stay if longer than 30 days

OTHER OUTCOMES:
Mortality | 6 months
Training induced enhancement of aerobic capacity : VO2 max, Endurance time, 6 MWT (m) | baseline, after the 4-6 week endurance training program (before surgery), and at 3 and 6 months follow-up
Health-related quality of life (SF-36) | at baseline and after the 4-6 week endurance training program(before surgery), and at 3 and 6 months follow-up
Analysis of the barriers for the use of communication and information technologies in prehabilitation program | Frame: 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Graciela Martinez Palli, Principal Investigator — Hospital Clinic de Barcelona, IDIBAPS
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Barberan-Garcia A, Ubre M, Pascual-Argente N, Risco R, Faner J, Balust J, Lacy AM, Puig-Junoy J, Roca J, Martinez-Palli G. Post-discharge impact and cost-consequence analysis of prehabilitation in high-risk patients undergoing major abdominal surgery: secondary results from a randomised controlled trial. Br J Anaesth. 2019 Oct;123(4):450-456. doi: 10.1016/j.bja.2019.05.032. Epub 2019 Jun 25. PMID 31248644